CLINICAL TRIAL: NCT03286387
Title: Contextual Associations During Episodic Recall of Everyday or Virtual Reality
Acronym: BREAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0404; 2017-A02558-45 (Other: ID-RCB)
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: Memory; naturalistic; context; fMRI; Attention
MeSH Terms: interventions — Functional Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Memory for naturalistic episodes (Experimental): Encoding of episode in real life situations (using Smartphones) or in a virtual environment, followed by memory retrieval (either behavior only or with fMRI, in successive studies)
  Interventions: Other: Functional brain imaging without any contrast agent

INTERVENTIONS:
Other: Functional brain imaging without any contrast agent — During the fMRI protocol, the subject will perform the retrieval tasks while whole-brain activity will be recorded using Echo Planar Imaging (EPI) that measures the Blood Oxygen Level Dependent (BOLD) signal (2x2x2 isotropic voxels, Echo Time (TE) = 30 ms, Repetition Time (TR) = 2.5 sec). The functional session will be subdivided into several parts ("Runs", duration: 10-15 min). Together with the functional data, the protocol will include a structural scan (T1 weighted, 1x1x1 mm voxels; duration 5-7 min) and a field mapping sequence (duration: 1 min).

SUMMARY:
The project is dedicated to development of new paradigms to investigate memory and attention in the rich and realistic environments. The investigator will use modern interactive digital technologies for encoding complex episodes either using mobile phone technology in everyday life or using a virtual reality life-like simulation.

He aims to characterize the role of the medial temporal lobe and prefrontal cortex during recall of naturalistic episodic experiences, using functional neuroimaging (fMRI) in healthy participants. The secondary aim is assess how the allocation of attention during memory encoding contribute to mechanisms of the subsequent recall. He will achieve this by monitoring gaze direction during encoding and by analyzing the retrieval data as a function of the elements that participants attended / fixated during encoding.

The protocol will involve, first, behavioral testing of memory performance with encoding in the real-life or in virtual reality, followed by the main hypothesis testing phase when fMRI will be used to measure brain activity during retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Possession a Smartphone compatible with GPS 3-rd generation and exploitation system Android 4.2 with user-activated geolocation (for mobile phone studies).
* Able to navigate in virtual reality with a help of the keyboard (for virtual reality studies).
* Not using glasses.
* All subjects will give their written consent for participation in the study.
* They will be right-handed
* They will have French social coverage.

Exclusion Criteria:

* Previous neurologic or psychiatric disease.
* Cognitive deficits restricting understanding of the tasks.
* Pregnant or breath-feeding women.
* Persons under guardianship, curatorship or any other administrative or judicial measure of deprivation of rights or liberty.
* Subjects currently participating in other study.

Additional exclusion criteria for an fMRI recording

* Neurologic, cardiac electrostimulation or defibrillator.
* Cardiac prostheses
* Intracranial clips or clamps
* Cerebrospinal fluid disorders
* Metal particles in the eyes
* Metal dental or articular prostheses
* Diffusion pomp or other infusion system
* Claustrophobia
* Head tattoo , makeup, hair gel

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
BOLD cerebral response to contextual recall in medial temporal lobe | up to 1 week after the end of the encoding session
  After spatial preprocessing of individual series of EPI fMRI images, normalization and smoothing as suggested for SPM analysis, the successful and failed contextual recall will be modeled and convolved with canonical HRF function. The GLM will be estimated according to the algorithm of SPM, the significance threshold will be p<0.05 FWE within the regions of interest. Our hypothesis will be confirmed by activation of medial temporal lobe and prefrontal cortex in contextual recall, congruent contextual cueing and recall of episodes when targets were semantically congruent with the context at encoding.
BOLD cerebral response to contextual recall in prefrontal cortex | up to 1 week after the end of the encoding session
  After spatial preprocessing of individual series of EPI fMRI images, normalization and smoothing as suggested for Statistical Parametric Mapping (SPM) analysis, the successful and failed contextual recall will be modeled and convolved with canonical HRF function. The GLM will be estimated according to the algorithm of SPM, the significance threshold will be p<0.05 Family-wise error (FWE) within the regions of interest. Our hypothesis will be confirmed by activation of medial temporal lobe and prefrontal cortex in contextual recall, congruent contextual cueing and recall of episodes when targets were semantically congruent with the context at encoding.

SECONDARY OUTCOMES:
Pattern of gaze fixation during episodic encoding and cerebral activity during recall | up to 1 week after the end of the encoding session
  The gaze direction during both during episodic encoding and recall. We will estimate a correlation between the activation of medial temporal lobe/ prefrontal cortex and the similarity of the gaze fixations during encoding and retrieval. A positive correlation will support our hypothesis about the link between attention and contextual encoding.

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano MACALUSO, PhD, Principal Investigator — INSERM U1028 - Impact - CRNL
Locations (1):
- U1028 INSERM - CNRS UMR 5292 Equipe ImpAct, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foudil SA, Macaluso E. The influence of the precuneus on the medial temporal cortex determines the subjective quality of memory during the retrieval of naturalistic episodes. Sci Rep. 2024 Apr 4;14(1):7943. doi: 10.1038/s41598-024-58298-y. PMID 38575698
- [Background] Foudil SA, Pleche C, Macaluso E. Memory for spatio-temporal contextual details during the retrieval of naturalistic episodes. Sci Rep. 2021 Jul 16;11(1):14577. doi: 10.1038/s41598-021-93960-9. PMID 34272405